CLINICAL TRIAL: NCT02382315
Title: Efficacy of a Cognitive-Existential Therapy Intervention to Address Fear of Recurrence in Men and Women With Cancer: A Randomized Clinical Trial
Brief Title: A Therapy Intervention to Address Fear of Recurrence in Men and Women With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20150013-01H
Record Dates: First submitted 2015-02-04; First posted 2015-03-06 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Cancer
Keywords: fear of cancer recurrence; psychosocial intervention; randomized controlled clinical trial
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): Fear of Cancer Recurrence Intervention.
  Interventions: Behavioral: Fear of Cancer Recurrence Intervention
- Wait-list Control Group (No Intervention): Patients assigned to this arm will be asked to wait 6 weeks before being offered the fear of cancer recurrence intervention.

INTERVENTIONS:
Behavioral: Fear of Cancer Recurrence Intervention — A 6-week individual therapy intervention to address fear of cancer recurrence in male and female cancer survivors. Patients will learn tools and techniques to help manage their fears, and learn to tolerate the uncertainty associated with the possibility of their cancer recurring.
  Arms: Intervention Group

SUMMARY:
Fear of cancer recurrence (FCR) is one of the most frequently cited unmet needs among survivors, and affects 22 to 87% of cancer patients. The objective of this study is to test the effectiveness of a six weekly, 1-hour manual-based individual therapy to reduce FCR among cancer survivors. A total of n=20 cancer survivors will be recruited from the Ottawa Hospital Cancer Centre (TOHCC) in Ottawa, Ontario. Participants will be randomly selected to receive either the psychotherapy intervention or standard care at TOHCC. All participants will be asked to complete a series of questionnaire packages at 3 time points. Ultimately, decreasing FCR can improve quality of life and reduce distress.The objective of this RCT study is to test the effectiveness of a six weekly, 1 hour manual-based cognitive-existential (CE) individual intervention to reduce FCR among cancer survivors. It is hypothesized that:

1. Participants in the intervention group will have lower scores on the primary outcome measure of FCR after treatment, as compared to a standard care control group
2. Participants in the intervention group will have lower scores on the secondary outcome measures of uncertainty, cancer-specific distress, intolerance of uncertainty, and faulty beliefs about worrying, will demonstrate enhanced coping skills, and report better quality of life after treatment, as compared to a standard care control group, and these changes will be maintained at a 3-month follow-up.

DETAILED DESCRIPTION:
Studies show that cancer survivors have a variety of unmet needs, with Fear of Cancer Recurrence (FCR) being the most frequently reported unmet need. FCR is defined as "the fear or worry that the cancer will return or progress in the same organ or in another part of the body", and has been described as the sword of Damocles that hangs over patients' heads for the rest of their lives. Up to 49% of survivors experience moderate-to-high FCR, with associated maladaptive coping such as hyper-vigilance, excessive bodily checking and reassurance seeking. There is clear evidence that a large portion of cancer survivors experience moderate-to-high FCR. There is a paucity of literature on psychosocial interventions that address FCR. To date, there is only one published intervention that has examined fear of disease progression, a concept related to FCR. Herschbach and colleagues examined the effects of a cognitive-behavioural group therapy and a supportive existential group therapy for patients with cancer or arthritis. Results indicated that both interventions successfully reduced fear of disease progression in patients when compared to a control group. However, the interventions were only effective for cancer patients. Humphris and Ozakinci developed the AFTER intervention to address FCR in head and neck cancer patients, although results of this study are yet to be published. Thewes and colleagues have developed and pilot-tested the Conquer Fear Intervention, which aims to address FCR in breast and colorectal cancer patients. This intervention is currently being evaluated in an RCT. As a result of the lack of published interventions and in order to address the needs of patients with moderate-to-high FCR, Lebel and Maheu designed a cognitive-existential group intervention to treat FCR. Lebel and colleagues adapted components of the intervention developed by Kissane and colleagues. The intervention consists of six consecutive, 1.5-hour weekly group therapy sessions, with homework exercises assigned each week. The authors pilot-tested the intervention with breast and ovarian cancer participants (n=44), and results of the study demonstrated significant improvement, with a moderate effect size between pre-and post-testing in FCR (0.73), cancer-specific distress (0.38), quality of life (0.54), uncertainty (0.41), and coping strategies (0.16-0.27). Almost all changes were sustained at 3-month follow-up. It appears that no individual therapeutic intervention exists for both men and women that specifically addresses FCR. The proposed study will address the gaps in the literature by adapting the aforementioned FCR group intervention to an individual therapy format.

The research design is a randomized controlled trial (RCT). This study is a two-arm, pre-post pilot study. Participants will be randomized into either an intervention arm or a wait-list control arm. Individuals randomized to the intervention arm will receive the six-week cognitive-existential intervention, and individuals randomized to the control arm will receive standard care at The Ottawa Hospital and be wait-listed for the intervention. Participants assigned to the control group will be informed at the beginning of the study that they will have the option to participate in the intervention after completing the control arm component (6 weeks later). Participants will be asked to complete a series of questionnaire packages. There will be 3 measurement occasions for participants randomized to the intervention group: one week prior to the intervention (during the pre-therapy meeting), one week after the end of the intervention, and 3 months following the end of the intervention. There will be 4 measurement occasions for participants randomized to the control group: 6 weeks prior to the intervention (during the pre-therapy meeting), immediately before the intervention begins, one week after the end of the intervention, and 3 months following the end of the intervention. Twenty (n=20) male and female cancer survivors from the greater Ottawa region will be recruited for the study. The aim is to recruit 10 males and 10 females from mixed cancer groups. Participants will be recruited from The Ottawa Hospital Cancer Centre (TOHCC). Participants will be recruited from TOHCC through personalized letters, by TOHCC circle of care staff members, through posting of study posters throughout TOHCC, by display of study posters at various cancer organizations (e.g., the Maplesoft Centre), and through use of OHRI's OBIEE tool. Individuals who are reached by personalized letter, by study posters, or through email will have the option to contact the research assistant via telephone for more information on the study. Participants who complete the patient information contact form will be asked to either return the form to their healthcare provider, or to place the form in the return box located in TOHCC waiting room. For individuals who complete the patient information contact form, the research assistant will collect the form and contact interested participants. Additionally, the investigators will use the OHRI's OBIEE tool to search for patients who have had a cancer diagnoses and have completed the TOH Consent to be Contacted for Research Purposes. The investigators will use the date range from January 2010-August 2014. The investigators will identify a pool of potential candidates for participation by requesting MOSAIC data from The Ottawa Hospital Cancer Centre. Once the investigators have this list of patients, they will screen the patient charts for eligibility to compile a list of potential participants who appear to be good candidates for the study. Patients who consented to be contacted for research may be contacted directly by a member of the research team or by their treating oncologist to inform about the study. Any patients for whom the investigators cannot find a signed consent to be contacted for research, a member of their circle of care (e.g., oncologist or nurse) will make the first contact and patients who are interested in learning more about the study and will then be contacted by the research coordinator. Participants will be screened for eligibility via telephone, and pre-therapy appointments will be set up should eligibility criteria be met. During the pre-therapy appointment, therapists will assess if participants are suitable for therapy, administer consent forms and the Mini-Mental State Examination, discuss general expectations, and prepare participants for the intervention. Once consent forms have been signed, participants will be assigned a participant number. All consent forms will be stored in a secured, locked room at the Ottawa Hospital, and will only be accessed by the research team. G*Power 3.1.5 was used to calculate the necessary sample size for a repeated measures ANOVA, between factors, with two groups (intervention group and standard care control group), and two measurement time points (pre- and post-intervention), using the effect size that was found in Lebel and colleagues' pilot study of 0.72 (φ=.80, p <.05). To obtain this effect size, a sample of 14 participants is required. While 14 participants is the minimum number to detect a difference between groups based on these parameters, approximately 20 participants will be recruited, in order to account for attrition.

Prior to randomization, the following forms will be completed for all eligible and consenting participants: 1) eligibility form 2) pre-therapy checklist and 3) consent form. Participants will be randomly assigned to one of the two study arms. Participants will first be stratified on gender prior to the randomization procedure, to ensure an equal number of men and women in both arms. Random assignment to each start time will be implemented via an online random number generator (http://www.randomizer.org) for the 20 participants. An individual with expertise on randomization outside of the research team will conduct the random assignment using this computerized procedure and keep the generated list, to ensure that participant assignment could not be identified by anyone on the research team. During the pre-therapy meeting, the consent forms will be explained to the participants. Once the consent forms are signed, participants will be asked to complete their first questionnaire package during the pre-therapy meeting. After completion of the questionnaire, the therapist will phone the aforementioned individual with the previously generated randomization list to find out which group the participant has been assigned to. The therapist will then inform the participants which group they were randomized to, and will then proceed to book the next appointment (i.e., either one week after if randomized to intervention group, or 6 weeks after if randomized to control group).Participants will be given the choice of completing online or paper-based questionnaires. Participants will be asked to complete the first questionnaire during the pre-therapy meeting. Participants randomized to the intervention arm will be informed of this outcome, and will schedule the first therapy session with their therapist for the following week.

Participants who prefer online questionnaires will be emailed the questionnaire packages via Fluid Survey, and will be asked to complete the questionnaires within 24 hours of receiving the survey email. Christina Tomei, Dr. Sophie Lebel, and Clinical Psychology doctoral students at the University of Ottawa will be the therapy facilitators. All therapy sessions will take place at the Ottawa Hospital's Psychosocial Oncology Program. Therapists will be asked to correspond and meet directly with their own clients. Clinical supervision will be provided for the therapy facilitators. All therapists will receive a one-day training under the direction of Christina Tomei and Dr. Sophie Lebel, who are well trained in the therapy. This approach to monitoring treatment integrity and fidelity has been successful in Lebel and colleagues' pilot study. All intervention sessions will be video-recorded, and reviewed independently by Dr. Sophie Lebel and Dr. Monique Lefebvre to assess treatment integrity and fidelity. The sessions will be rated for adherence to the content of the intervention using a 1-10 point Likert scale. Rating scales will be used to measure adherence to content (1-10), adequate processing of affect (1-10), and efficient time management (1-10). If adherence is less than 80% on any of these scales, additional over-the-telephone feedback will be provided. To maximize attendance, participants will be told about the importance of attending all six sessions at the time informed consent is to be obtained. For participants who miss more than one session, they will be asked to withdraw from the study, as too much material will have been missed. Participants will also be reimbursed for their travel expenses for each session. If participants choose to withdraw from the study, they can terminate without any consequence. Reasons for termination will be documented. Participants who select the online questionnaire option will be assigned a participant number, and will be provided with a link to complete their questionnaire package via Fluid Survey, and will receive reminder emails to complete their questionnaires. Participants who select the paper-based option will also be assigned a participant number, and will have questionnaire packages mailed to them at each respective measurement timepoint. Total completion time of each questionnaire package should take 20-30 minutes. A pre-post test design with a control group will be used. In order to examine treatment gains over time, several repeated-measures ANOVAs will be conducted, using a Bonferroni correction to adjust for multiple comparisons. The independent variable will have two-levels: time (pre-treatment and post-treatment), and treatment type (intervention versus standard care). The dependent variables will be FCR, quality of life, intolerance of uncertainty, reassurance seeking, impact of events, cancer-specific distress, beliefs about benefits of worrying, and coping. An intent-to-treat approach will be used: participants who drop out will be asked to complete their questionnaires and will be kept in the final analyses. Risks are minimal, but it is possible that a participant may not benefit from the intervention and may experience heightened anxiety during his or her participation in the program. Therapy facilitators will be responsible for providing referrals for individual counselling within the Psychosocial Oncology Program, should participants require additional resources. Additionally, the strictest confidentiality will be ensured when storing participant data. Participants will be informed that their participation in the study will be documented electronically on their hospital chart (i.e., vOACIS). Participants will be informed that notice of their involvement in the study will be accessible to members of The Ottawa Hospital team who have worked with them (e.g., physician, nurse). Participants will be informed that all identifying information and questionnaires will be kept in a secured, locked location at The Ottawa Hospital. This information will be kept in a separate password-protected electronic file. The proposed research has direct implications for clinical services development to improve quality of life for patients with cancer. Based on Lebel and colleagues' pilot data, it is possible that this RCT can demonstrate the effectiveness of this new psychosocial intervention to improve FCR and psychological functioning following treatment. Ultimately, this intervention may help women and men with elevated levels of FCR, and can result in improved coping and improve and restore quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Men and women diagnosed with cancer (stages I-III),
* English-speaking,
* 18 years of age or older,
* clinical level of FCR as indicated by a score of 13 or greater on the severity subscale of the FCRI (range 0-36),
* clinical distress score as indicated by a score of at least 24 on the IES (range 0-75),
* completion of cancer treatment,
* current or previous patients of the Ottawa Hospital Cancer Centre.

Exclusion Criteria:

* the refusal to provide informed consent,
* non-understanding of the English language,
* Stage IV cancer,
* previous cancer recurrence,
* currently enrolled in psychotherapy for cancer issues (whether individual or group) during the treatment,
* self-disclosure of unmanaged mental health disorder,
* have not been a patient of the Ottawa Hospital Cancer Centre.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-03; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Fear of Cancer Recurrence Inventory | Up to 7 Months
  The Fear of Cancer Recurrence Inventory (FCRI; Simard & Savard, 2009) is a 42-item multidimensional instrument that has been used to examine FCR

SECONDARY OUTCOMES:
The Impact of Events Scale | Up to 7 Months
  The Impact of Events Scale (IES; Horowitz, Wilner, & Alvarez, 1979) is a 15-item scale that measures the frequency of intrusive and avoidant thoughts associated with cancer
Perceived Risk of Cancer Recurrence | Up to 6 Months
  Perceived Risk of Cancer Recurrence will be measured using Bish, Sutton, Jacobs, Levine, Ramirez, & Hodgson's (2002) one-item measure. The question asks participants to rate their perceived risk of cancer recurrence relative to other people their age over the past two days.
The SF-8 Health Survey | Up to 7 Months
  The SF-8 Health Survey (Ware, Kosinski, Dewey, & Gandek, 2001) will be used to measure quality of life. The SF-8 is an eight-item health-related quality of life measure that provides an assessment of eight domains within a four-week recall period.
The Intolerance of Uncertainty Scale | Up to 7 Months
  The Intolerance of Uncertainty Scale (IUS; original French version: Freeston, Rheaume, Letarte, Dugas, & Ladouceur, 1994, English version: Buhr & Dugas, 2002) is a 27-item self-report measure that assesses individuals' beliefs about uncertainty.
The Mishel Uncertainty in Illness Scale - Community form | Up to 7 Months
  The Mishel Uncertainty in Illness Scale - Community form (MUIS-C) is a 23-item self-report measure that examines uncertainty in relation to diagnosis, treatment, and planning for the future in patients with cancer
The Cognitive Avoidance Questionnaire | Up to 7 Months
  The Cognitive Avoidance Questionnaire (CAQ; original French version: Gosselin, Langlois, Freeston, Ladouceur, Dugas, & Pelletier, 2002, English version: Sexton & Dugas, 2008) will be used to measure coping. The CAQ is a 25-item self-report measure that assesses the tendency to employ cognitive avoidance strategies when encountering intrusive thoughts (Sexton & Dugas, 2008)
The Health Anxiety Questionnaire: Reassurance-seeking behaviours subscale | Up to 7 Months
  The Health Anxiety Questionnaire Reassurance-seeking behaviours subscale (HAQ, Lucock & Morley, 1996) will be used to measure coping. This subscale consists of three items that pertain to body-checking and reassurance-seeking from loved ones over the course of the week.
The Reassurance Questionnaire | Up to 7 Months
  The Reassurance Questionnaire (RQ; Speckens, Spinhoven, Van Hemert, & Bolk, 2000) will be used to measure coping. The RQ is a 10-item self-report questionnaire that assesses the extent to which individuals feel reassured by their physician.

CONTACTS AND LOCATIONS:
Overall Officials: Monique Lefebvre, Ph.D., Principal Investigator — The Ottawa Hospital

REFERENCES:
- [Background] Armes J, Crowe M, Colbourne L, Morgan H, Murrells T, Oakley C, Palmer N, Ream E, Young A, Richardson A. Patients' supportive care needs beyond the end of cancer treatment: a prospective, longitudinal survey. J Clin Oncol. 2009 Dec 20;27(36):6172-9. doi: 10.1200/JCO.2009.22.5151. Epub 2009 Nov 2. PMID 19884548
- [Background] Baker F, Denniston M, Smith T, West MM. Adult cancer survivors: how are they faring? Cancer. 2005 Dec 1;104(11 Suppl):2565-76. doi: 10.1002/cncr.21488. PMID 16258929
- [Background] Butow PN, Bell ML, Smith AB, Fardell JE, Thewes B, Turner J, Gilchrist J, Beith J, Girgis A, Sharpe L, Shih S, Mihalopoulos C; members of the Conquer Fear Authorship Group. Conquer fear: protocol of a randomised controlled trial of a psychological intervention to reduce fear of cancer recurrence. BMC Cancer. 2013 Apr 23;13:201. doi: 10.1186/1471-2407-13-201. PMID 23617696
- [Background] Glynne-Jones R, Chait I, Thomas SF. When and how to discharge cancer survivors in long term remission from follow-up: the effectiveness of a contract. Clin Oncol (R Coll Radiol). 1997;9(1):25-9. doi: 10.1016/s0936-6555(97)80055-6. PMID 9039810
- [Background] Gupta SK. Intention-to-treat concept: A review. Perspect Clin Res. 2011 Jul;2(3):109-12. doi: 10.4103/2229-3485.83221. PMID 21897887
- [Background] Hart SL, Latini DM, Cowan JE, Carroll PR; CaPSURE Investigators. Fear of recurrence, treatment satisfaction, and quality of life after radical prostatectomy for prostate cancer. Support Care Cancer. 2008 Feb;16(2):161-9. doi: 10.1007/s00520-007-0296-x. Epub 2007 Jul 19. PMID 17638026
- [Background] Herschbach P, Keller M, Knight L, Brandl T, Huber B, Henrich G, Marten-Mittag B. Psychological problems of cancer patients: a cancer distress screening with a cancer-specific questionnaire. Br J Cancer. 2004 Aug 2;91(3):504-11. doi: 10.1038/sj.bjc.6601986. PMID 15238979
- [Background] Herschbach P, Berg P, Waadt S, Duran G, Engst-Hastreiter U, Henrich G, Book K, Dinkel A. Group psychotherapy of dysfunctional fear of progression in patients with chronic arthritis or cancer. Psychother Psychosom. 2010;79(1):31-8. doi: 10.1159/000254903. Epub 2009 Nov 4. PMID 19887889
- [Background] Horowitz M, Wilner N, Alvarez W. Impact of Event Scale: a measure of subjective stress. Psychosom Med. 1979 May;41(3):209-18. doi: 10.1097/00006842-197905000-00004. PMID 472086
- [Background] Humphris G, Ozakinci G. The AFTER intervention: a structured psychological approach to reduce fears of recurrence in patients with head and neck cancer. Br J Health Psychol. 2008 May;13(Pt 2):223-30. doi: 10.1348/135910708X283751. PMID 18492319
- [Background] Kissane DW, Bloch S, Miach P, Smith GC, Seddon A, Keks N. Cognitive-existential group therapy for patients with primary breast cancer--techniques and themes. Psychooncology. 1997 Mar;6(1):25-33. doi: 10.1002/(SICI)1099-1611(199703)6:13.0.CO;2-N. PMID 9126713
- [Background] Kissane DW, Bloch S, Smith GC, Miach P, Clarke DM, Ikin J, Love A, Ranieri N, McKenzie D. Cognitive-existential group psychotherapy for women with primary breast cancer: a randomised controlled trial. Psychooncology. 2003 Sep;12(6):532-46. doi: 10.1002/pon.683. PMID 12923794
- [Background] Ladouceur R, Dugas MJ, Freeston MH, Leger E, Gagnon F, Thibodeau N. Efficacy of a cognitive-behavioral treatment for generalized anxiety disorder: evaluation in a controlled clinical trial. J Consult Clin Psychol. 2000 Dec;68(6):957-64. PMID 11142548
- [Background] Lebel S, Rosberger Z, Edgar L, Devins GM. Comparison of four common stressors across the breast cancer trajectory. J Psychosom Res. 2007 Sep;63(3):225-32. doi: 10.1016/j.jpsychores.2007.02.002. Epub 2007 Aug 2. PMID 17719358
- [Background] Lebel, S. & Maheu. C. (2009). Development of a cognitive-existential intervention to address fear of cancer recurrence in women with cancer. Unpublished manuscript.
- [Background] Lebel S, Tomei C, Feldstain A, Beattie S, McCallum M. Does fear of cancer recurrence predict cancer survivors' health care use? Support Care Cancer. 2013 Mar;21(3):901-6. doi: 10.1007/s00520-012-1685-3. Epub 2012 Dec 27. PMID 23269420
- [Background] Lebel S, Maheu C, Lefebvre M, Secord S, Courbasson C, Singh M, Jolicoeur L, Benea A, Harris C, Fung MF, Rosberger Z, Catton P. Addressing fear of cancer recurrence among women with cancer: a feasibility and preliminary outcome study. J Cancer Surviv. 2014 Sep;8(3):485-96. doi: 10.1007/s11764-014-0357-3. Epub 2014 Apr 23. PMID 24756313
- [Background] Lee-Jones C, Humphris G, Dixon R, Hatcher MB. Fear of cancer recurrence--a literature review and proposed cognitive formulation to explain exacerbation of recurrence fears. Psychooncology. 1997 Jun;6(2):95-105. doi: 10.1002/(SICI)1099-1611(199706)6:23.0.CO;2-B. PMID 9205967
- [Background] Llewellyn CD, Weinman J, McGurk M, Humphris G. Can we predict which head and neck cancer survivors develop fears of recurrence? J Psychosom Res. 2008 Dec;65(6):525-32. doi: 10.1016/j.jpsychores.2008.03.014. Epub 2008 Sep 24. PMID 19027440
- [Background] Lucock, M. P., & Morley, S. (1996). The health anxiety questionnaire. British Journal of Health Psychology, 1(2), 137-150. doi: 10.1111/j.2044-8287.1996.tb00498.x
- [Background] Mishel MH. The measurement of uncertainty in illness. Nurs Res. 1981 Sep-Oct;30(5):258-63. PMID 6912987
- [Background] Muzzin LJ, Anderson NJ, Figueredo AT, Gudelis SO. The experience of cancer. Soc Sci Med. 1994 May;38(9):1201-8. doi: 10.1016/0277-9536(94)90185-6. PMID 8016685
- [Background] Savard J, Ivers H. The evolution of fear of cancer recurrence during the cancer care trajectory and its relationship with cancer characteristics. J Psychosom Res. 2013 Apr;74(4):354-60. doi: 10.1016/j.jpsychores.2012.12.013. Epub 2013 Jan 26. PMID 23497839
- [Background] Sexton KA, Dugas MJ. The Cognitive Avoidance Questionnaire: validation of the English translation. J Anxiety Disord. 2008;22(3):355-70. doi: 10.1016/j.janxdis.2007.04.005. Epub 2007 Apr 25. PMID 17544253
- [Background] Simard S, Savard J. Fear of Cancer Recurrence Inventory: development and initial validation of a multidimensional measure of fear of cancer recurrence. Support Care Cancer. 2009 Mar;17(3):241-51. doi: 10.1007/s00520-008-0444-y. Epub 2008 Apr 15. PMID 18414902
- [Background] Simard S, Savard J, Ivers H. Fear of cancer recurrence: specific profiles and nature of intrusive thoughts. J Cancer Surviv. 2010 Dec;4(4):361-71. doi: 10.1007/s11764-010-0136-8. Epub 2010 Jul 10. PMID 20617394
- [Background] Simard S, Thewes B, Humphris G, Dixon M, Hayden C, Mireskandari S, Ozakinci G. Fear of cancer recurrence in adult cancer survivors: a systematic review of quantitative studies. J Cancer Surviv. 2013 Sep;7(3):300-22. doi: 10.1007/s11764-013-0272-z. Epub 2013 Mar 10. PMID 23475398
- [Background] Speckens AEM, Spinhoven P, Van Hemert AM, Bolk JH. The Reassurance Questionnaire (RQ): psychometric properties of a self-report questionnaire to assess reassurability. Psychol Med. 2000 Jul;30(4):841-7. doi: 10.1017/s0033291799002378. PMID 11037092
- [Background] Thewes B, Butow P, Bell ML, Beith J, Stuart-Harris R, Grossi M, Capp A, Dalley D; FCR Study Advisory Committee. Fear of cancer recurrence in young women with a history of early-stage breast cancer: a cross-sectional study of prevalence and association with health behaviours. Support Care Cancer. 2012 Nov;20(11):2651-9. doi: 10.1007/s00520-011-1371-x. Epub 2012 Feb 11. PMID 22328003
- [Background] Thewes B, Butow P, Zachariae R, Christensen S, Simard S, Gotay C. Fear of cancer recurrence: a systematic literature review of self-report measures. Psychooncology. 2012 Jun;21(6):571-87. doi: 10.1002/pon.2070. Epub 2011 Oct 21. PMID 22021099
- [Background] Urbaniak, G. C., & Plous, S. (2007). Research randomizer. Retrieved from http://www.randomizer.org
- [Background] Vickberg SM. The Concerns About Recurrence Scale (CARS): a systematic measure of women's fears about the possibility of breast cancer recurrence. Ann Behav Med. 2003 Winter;25(1):16-24. doi: 10.1207/S15324796ABM2501_03. PMID 12581932